CLINICAL TRIAL: NCT03386370
Title: Indian Registry (The INDigo System in Acute Lower Limb malperfusioN)
Brief Title: The Indigo System in Acute Lower Limb Malperfusion
Acronym: INDIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Responsible Party: Principal Investigator, Carlo Setacci, Gianmarco de Donato, University of Siena, Azienda Ospedaliera Universitaria Senese
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Indian001
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Acute Ischemia of Lower Limb
Keywords: Acute ischemia; Lower Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment by "Indigo" mechanical thrombectomy system (Other): Acute or Chronic clot: if chronic (> 14 days) no intervention given via Indigo
  Interventions: Device: "Indigo" Mechanical Thrombectomy System

INTERVENTIONS:
Device: "Indigo" Mechanical Thrombectomy System — Removal of acute clot (< 14 days) from the artery causing lower limb ischemia, using the "Indigo" System by Penumbra

SUMMARY:
To evaluate, in a controlled setting, the early safety and effectiveness of the Penumbra/Indigo aspiration thrombectomy Systems (San Francisco, California), and to define optimal technique for the use of these systems in patients with confirmed peripheral acute occlusions.

ELIGIBILITY:
Patients will be selected based on the investigator's assessment and evaluation of the underlying disease.

The patient's medical condition should be stable, with no underlying medical condition that would prevent them from performing the required testing or from completing the study.

Patients should be geographically stable, willing and able to cooperate in this clinical study, and remain available for mid term follow-up. Patients who do not wish to participate in this study can obtain any other standard commercially available device therapy. Refusal to participate in this study will in no way affect their care at the institution.

Inclusion Criteria

* Patient presenting with an acute occlusion of lower limb arteries (thrombosis no longer than 14 days)
* Patient presenting a score from I to IIb following Rutherford classification for acute limb ischemia
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient is eligible for treatment with the Indigo System (Penumbra)

Exclusion Criteria

* Estimated time of intraluminal thrombus > 14 days
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients with a history of prior life-threatening contrast medium reaction
* Life expectancy of less than six months
* Any patient considered to be hemodynamically unstable at onset of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Technical success of the thromboaspiration with the Indigo system. | At intra-procedural completion angiography
  The primary endpoint of the study is the technical success of the thromboaspiration with the Indigo system. Assessment of vessel patency will be recorded using the Thrombolysis in Myocardial Infarction (TIMI) score classifications both before and after use of the device.

SECONDARY OUTCOMES:
Clinical success at 1 month follow-up. | 1 month
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Safety Rate at discharge: Serious adverse event. | 1 month
  Safety rate at discharge, defined as absence of any serious adverse events (SAE). A SAE is defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability.
Primary Patency | 1 month
  Primary patency at 1 month. Primary patency is defined as a target lesion without a hemodynamically significant stenosis/reocclusion on duplex ultrasound (>50%,) and without target lesion reintervention (TLR) within 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular Surgery, University of Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamada R, Adams J, Guimaraes M, Schonholz C. Advantages to Indigo mechanical thrombectomy for ALI: device and technique. J Cardiovasc Surg (Torino). 2015 Jun;56(3):393-400. Epub 2015 Feb 3. PMID 25644826